**Cover Page** 

Title: A Prospective Study of Evaluation of Operative Duration as a Predictor of Mortality in

Pediatric Emergency Surgery: Concept of 100 Minutes Laparotomy in Resource-limited

Setting

NCT Identifier Number: Not assigned

**Document Date:** 31/03/2017

**Informed Consent for Participation in Study** 

My child was brought by me in the casualty of JN Medical College and Hospital on date

. He/she was managed appropriately and in timely manner to the best of my

knowledge. He/she was then operated under my due informed consent in the emergency

operation theatre of the hospital by Dr Kaushal Deep Singh. The effect and nature of operation

and anaesthesia and associated risks were explained to me by the above mentioned operating

surgeon. I was told about this study which is being undertaken at the hospital and strongly

believe that this is not a trial and error experiment; rather a manner of scientific and appropriate

gathering of data being done to improve final patient outcome. I agree to get my ward to be

part of this study at Jawaharlal Nehru Medical College, Aligarh Muslim University, Aligarh.

Signature of Patient's Parent/Guardian:

Date of Consent:

Consent verified by (Name, Designation and Signature):